CLINICAL TRIAL: NCT06602726
Title: A Randomized, Double-masked, Placebo-controlled Study to Assess the Efficacy and Safety of REGN1908-1909 to Reduce Signs and Symptoms of Allergic Conjunctivitis in Participants With Cat Allergy
Brief Title: A Study to Demonstrate How Well REGN1908-1909 Works in Reducing Ocular Allergy Signs and Symptoms in Adult Participants With Cat Allergy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R1908-1909-ALG-2416
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Allergic Conjunctivitis
Keywords: Cat allergy; Eye allergy; Ocular allergy; Ocular allergy symptoms; Ocular allergy signs
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- REGN1908-1909 (Experimental)
  Interventions: Drug: REGN1908; Drug: REGN1909
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REGN1908 — Administered per the protocol
  Arms: REGN1908-1909
Drug: REGN1909 — Administered per the protocol
  Arms: REGN1908-1909
Drug: Placebo — Administered per the protocol
  Arms: Placebo

SUMMARY:
This study is researching 2 experimental drugs, REGN1908 and REGN1909, which are called REGN1908-1909 when mixed together (called "study drug") to reduce eye allergy signs and symptoms from cat allergy.

The aim of the study is to see how safe and effective the study drug is at lowering allergic eye signs and symptoms compared with placebo. A placebo looks like a treatment but does not contain any real medicine.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Documented or participant-reported history of moderate to severe cat allergy for at least 2 years with bothersome ocular symptoms being near cat(s)
2. Positive SPT with cat allergen extract (mean wheal diameter at least 5 mm greater than the negative control) at screening visit 1
3. Positive Allergen-specific Immunoglobulin E (sIgE) tests for cat allergen and Fel d 1 (both ≥0.7 kUa/L) at screening visit 1
4. Must be able to complete the screening CACs to confirm moderate to severe cat allergen-induced allergic conjunctivitis as described in the protocol
5. Must not have lived with a cat(s) in the home for the past 3 years and must be willing to have no exposure to cat(s) at home throughout the study duration as described in the protocol

Key Exclusion Criteria:

1. Participation in a prior clinical study and received either REGN1908-1909, REGN1908, or REGN1909 antibodies as described in the protocol
2. Inability to complete or termination of the screening or confirmatory CAC (where applicable) due to a safety concern (eg, anaphylaxis), per PI judgement
3. Significant and/or severe allergies, ocular, nasal, or systemic disease causing symptoms (eg, ocular itching, ocular redness, etc) that are expected to coincide or potentially interfere with the study CAC assessments, as described in the protocol
4. Persistent chronic or recurring acute infection requiring treatment with systemic antibiotics, antivirals, or antifungals, or any untreated respiratory infections within 4 weeks prior to screening visit 1 as described in the protocol
5. Presence of ocular conditions associated with acute or chronic vision loss, or any other ophthalmic disease or abnormality that may affect the study outcomes or participant safety, per Principal Investigator (PI) judgement as described in the protocol
6. Uncontrolled asthma or on Global Initiative for Asthma (GINA) steps 4 to 5 as described in the protocol
7. Abnormal lung function as judged by the investigator with Forced expiratory volume in 1 second (FEV1) <70% of predicted at screening
8. History of cat immunotherapy (eg, subcutaneous immunotherapy or any other route) in the 3 years prior to screening visit 1
9. Ongoing Allergen immunotherapy (AIT) with any allergen other than cat at screening visit 1 as described in the protocol

Note: Other Protocol Defined Inclusion/ Exclusion Criteria Apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-08-02 (Actual)

PRIMARY OUTCOMES:
Ocular itch score | At day 8 post-Conjunctival Allergen Challenge (CAC)
  Assessed using the Ora Calibra® Conjunctival Allergen Challenge Ocular Itching Scale, a 0-4 point scale where 0= none and 4= incapacitating itch, 0.5 unit increments

SECONDARY OUTCOMES:
Conjunctival redness score | At day 8 post-CAC
  Assessed using the Ora Calibra® Hyperemia Scale (for conjunctival [conjunctival redness scale], ciliary [ciliary redness scale] and episcleral [episcleral redness scale] vessel beds), a 0 to 4 point scale, where 0 = none and 4 = extremely severe, 0.5 unit increments
Percent change in cat titrated Skin prick test (tSPT) | Baseline and day 8
  Area under the curve (AUC) of the mean wheal diameters
Tearing score | At day 8 post-CAC
  Assessed using the Ora Calibra® Conjunctival Allergen Challenge Tearing Scale, a 0-4 scale where 0 = none and 4 = very severe, 1 unit increments
Total Ocular Symptom Score (TOSS) | At day 8 post-CAC
  TOSS is a summed score of ocular itch score (graded 0 = none to 4 = incapacitating itch), conjunctival redness score (graded 0 = none to 4 = extremely severe), and tearing score (graded 0 = none to 4 = very severe) for a total range from 0 to 12, where higher scores indicate worse responses
Total redness score | At day 8 post-CAC
  The total redness score is calculated for CAC: range 0 to 12, where higher scores indicate worse responses (calculated as a sum of the bilateral averages for conjunctival redness score, graded 0 = none to 4 = extremely severe + ciliary redness score, graded 0 = none and 4 = extremely severe + episcleral redness score, graded 0 = none and 4 = extremely severe)
Ciliary redness score | At day 8 post-CAC
  Assessed using the Ora Calibra® Hyperemia Scale (for conjunctival [conjunctival redness scale], ciliary [ciliary redness scale] and episcleral [episcleral redness scale] vessel beds), a 0 to 4 point scale, where 0 = none and 4 = extremely severe, 0.5 unit increments
Episcleral redness score | At day 8 post-CAC
  Assessed using the Ora Calibra® Hyperemia Scale (for conjunctival [conjunctival redness scale], ciliary [ciliary redness scale] and episcleral [episcleral redness scale] vessel beds), a 0 to 4 point scale, where 0 = none and 4 = extremely severe, 0.5 unit increments
Change in cat tSPT | Baseline and day 8
  AUC of the mean wheal diameters
Change in cat tSPT | Baseline and day 113
  AUC of the mean wheal diameters
Percent change in cat tSPT | Baseline and day 113
  AUC of the mean wheal diameters
Incidence of Treatment-emergent adverse events (TEAEs) | Up to Day 113
Severity of TEAEs | Up to Day 113
Incidence of serious TEAEs | Up to Day 113
Incidence of Adverse event of special interest (AESIs) | Up to Day 113
Total REGN1908 concentrations in serum over time | Up to Day 113
Total REGN1909 concentrations in serum over time | Up to Day 113
Incidence of Anti-drug antibodies (ADAs) to REGN1908 | Up to Day 113
Titers of ADAs to REGN1908 | Up to Day 113
Incidence of ADAs to REGN1909 | Up to Day 113
Titers of ADAs to REGN1909 | Up to Day 113

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (4):
- Andover Eye Associates, Andover, Massachusetts, United States
- Canada (3):
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Red Maple Trials Inc., Ottawa, Ontario
  - Clinique de Specialisee en Allergie de la Capitale, Québec

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/